CLINICAL TRIAL: NCT01728974
Title: Mechanisms of Pharyngeal Collapse in Sleep Apnea
Brief Title: Mechanisms of Pharyngeal Collapse in Sleep Apnea, Study A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Andrew Wellman, Andrew Wellman, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012P000957A; 1R01HL102321-01A1 (NIH)
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Obstructive Sleep Apnea; Pathophysiology
Keywords: Obstructive Sleep Apnea; Pathophysiology
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharyngeal topical anesthesia (Experimental): Pharyngeal topical anesthesia will be performed using 4% lidocaine spray
  Interventions: Other: Pharyngeal topical anesthesia

INTERVENTIONS:
Other: Pharyngeal topical anesthesia — Pharyngeal topical anesthesia will be performed using 4% lidocaine spray

SUMMARY:
In obstructive sleep apnea, the upper airway recurrently closes during sleep. The mechanisms that lead to airway closure are not completely understood. While the airway of some people narrows and airflow decreases during inspiration due to increasing inspiratory effort, others maintain constant airflow throughout inspiration. Airway neuromuscular reflexes may protect against airway narrowing that occurs due to increasing inspiratory effort. To test this hypothesis, the investigators will initially measure airway neuromuscular reflex and inspiratory flow and then attenuate neuromuscular reflex through topical pharyngeal anesthesia to observe the effects on inspiratory flow.

DETAILED DESCRIPTION:
The mechanisms that lead to airway closure are not completely understood. While the airway of some people narrows and airflow decreases during inspiration due to increasing inspiratory effort, others maintain constant airflow throughout inspiration (negative effort dependence, NED). The investigators hypothesize that upper airway neuromuscular reflexes may protect against narrowing that occurs due to increasing inspiratory effort. Topical oropharyngeal anesthesia has been shown to reduce neuromuscular reflexes. Thus, the investigators also hypothesize that patients with stable inspiratory flow will develop NED once the reflexes have been impaired with topical anesthetic. The investigators plan to:

1. measure upper airway muscle EMG to assess how it corresponds to the presence or absence of NED. This aim will allow us to test the hypothesis that robust upper airway muscle reflexes can protect against NED.
2. reduce upper airway muscle activity and reflexes by topical oropharyngeal anesthesia. This will allow us to test the hypothesis that attenuated upper airway muscle activity induced by topical anesthesia can induce NED.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects or patients with OSA

Exclusion Criteria:

* Any unstable cardiac condition (other than well controlled hypertension) or pulmonary problems.
* Any medication known to influence breathing, sleep/arousal or muscle physiology
* Concurrent sleep disorders (insomnia, narcolepsy, central sleep apnea or parasomnia)
* Claustrophobia
* Inability to sleep supine
* Allergy to lidocaine or oxymetazoline HCl
* For women: Pregnancy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-12-08 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Negative effort dependence variation | After pharyngeal topical anesthesia
  The magnitude of negative effort dependence will be expressed as the percent decrease in inspiratory flow from Vmax. NED will be compared before and after topical upper airway anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: David A Wellman, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States